CLINICAL TRIAL: NCT05253534
Title: Pilot Study to Evaluate Clinically the Short-Term Efficacy of GlaucoT Glaucoma Treatment Glasses in the Treatment of Primary Open-Angle Glaucoma (GlaucoT)
Brief Title: GlaucoT Glaucoma Treatment Glasses in the Treatment of Primary Open-Angle Glaucoma
Acronym: GlaucoT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaucot Teknoloji Anonim Sirketi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-169
Record Dates: First submitted 2022-02-02; First posted 2022-02-23 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Primary Open-Angle Glaucoma
Keywords: Glaucoma; Neuroprotection; Gamma Rhythm; Non-invasive; Wearable
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Intervention Model Description: Evaluation of the efficacy and safety of GlaucoT in patients with primary open-angle glaucoma (POAG)
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- Gamma Rhythm Stimulation Group (Experimental): Evaluation of the efficacy and safety of GlaucoT in patients with primary open-angle glaucoma (POAG).
  In this study, it was planned to investigate the effect of reducing the progression of glaucomatous damage by applying 40 Hz flicker light therapy for 1 hour a day to POAG patients. It is planned to use visual field test, measurements of retinal nerve fiber layer (RNFL) and ganglion cell complex (GCC) layer thicknesses in optical coherence tomography to investigate the effectiveness of the treatment.
  Interventions: Device: GlaucoT Glaucoma Treatment Device
- Control Group (No Intervention): This group will be monitored without using the device.The data will be used only for comparison.
  Considering the sample size calculations and losses, a total of 60 patients are planned to be included in the study, with 30 patients in each group.

INTERVENTIONS:
Device: GlaucoT Glaucoma Treatment Device — In this study, flicker light therapy, the effectiveness of which was investigated in the treatment of glaucoma based on some methods used in different diseases, is described for the first time in glaucoma.
  Studies investigating the neurodegenerative properties of glaucoma have found similarities in the pathophysiology of Alzheimer's disease and glaucoma.
  40 Hz flicker of light Alzheimer 's the positive effects on the knitted cortex have also been shown in studies. 40 Hz flicker light is aimed to reduce glaucoma and retinal ganglion cell loss due to glaucoma, by reducing neurodegeneration by decreasing amyloid and metabolite accumulation by increasing both microglial phagocytic activation effect and retinal blood flow.
  Arms: Gamma Rhythm Stimulation Group

SUMMARY:
Glaucoma is a chronic and progressive optic neuropathy characterized by degeneration of ganglion cells and axons with loss of visual function.

It is estimated that glaucoma, which is the second cause of preventable blindness in the world, affects nearly 60 million people worldwide.

The most common type of glaucoma is primary open-angle glaucoma (POAG). POAG is a chronic progressive optic neuropathy with characteristic morphological changes in the optic nerve head and retinal nerve fiber.

POAG, progressive retinal ganglion cell death and visual field loss are associated with these changes.

Risk factors for POAG are age, race, high intraocular pressure (IOP), family history of glaucoma, thin central corneal thickness (CCT), high myopia. IOP is the only modifiable risk factor that we can control. For this reason, the priority in the treatment of POAG has always been to reduce IOP. In glaucoma, the essential point is to preserve the damaged ganglion cell layer and therefore the visual functions. In addition to clinical examination, visual field measurements that measure functions, optical coherence tomography (OCT) thickness measurements that measure anatomical changes, and optic nerve head parameters are the most reliable methods for both diagnosis and evaluation of the efficacy of treatment.

Following the results of the visual field and OCT measurements, it will be tried to determine to what extent glaucoma damage can be ceased by the developed GlaucoT glaucoma treatment glasses.

In this study, it is aimed to measure the effectiveness and safety of flicker light therapy, the effectiveness of which has been investigated in the treatment of Alzheimer's previously and has clinically significant results, with the GlaucoT glaucoma treatment glasses, which was developed to cease visual field loss with patient comfort at the forefront and at a lower cost.

DETAILED DESCRIPTION:
Background:

Glaucoma, a neurodegenerative disease, is characterized by the death of retinal ganglion cells and their axons. This damage affects all visual pathways up to the visual center in the brain.

Although increased intraocular pressure is considered the most important modifiable risk factor in glaucoma, many factors play a role in its pathogenesis and progression.

Different classifications have been proposed for various types of glaucoma. Accordingly, glaucoma;

* Open angle or closed angle depending on the iridocorneal angle,
* Primary or secondary, depending on the presence of etiological factors that may cause increased intraocular pressure,
* According to the age of onset of glaucoma, it can be classified as congenital, childhood or adult glaucoma.

In general, POAG is the most common type of glaucoma, accounting for 60-70% of cases. This is followed by secondary glaucomas (30%), primary angle-closure glaucomas (12%) and congenital glaucomas (3%).

POAG, also known as simple chronic glaucoma, is a disease with elevated intraocular pressure, cupping at the optic nerve head, and loss of visual field.

POAG is an insidious onset, progressive, bilateral anterior optic neuropathy. One of the features that distinguishes it from other types of glaucoma is the open appearance of the iridocorneal angle.

The most common type of glaucoma is POAG, and its incidence is 0.5-6.6% over the age of 40 in western countries. The incidence of POAG increases with age.

POAG is a progressive neurodegenerative optic neuropathy characterized by high IOP (≥21 mmHg), glaucomatous optic disc, retinal ganglion cells and retinal nerve fiber layer (RNFL) damage, and open iridocorneal angle.

POAG is bilateral and usually has an asymmetrical onset. Until the last period, it usually does not give any symptoms.

POAG is the most common type of open-angle glaucoma and is one of the leading causes of preventable blindness. Since POAG is asymptomatic in the early stages, the diagnosis is usually made after irreversible visual damage has occurred. With early diagnosis and appropriate treatment, the disease can be caught before significant loss of vision develops.

Open iridocorneal angle, IOP above 21 mm Hg, and vertical enlargement of the optic disc cupping are clinical findings of POAG.

As a result of the glaucomatous damage, severe visual field and visual acuity losses develop.

Although the biggest risk factor for the progression of the disease is high IOP, it is known that other factors also play a role, and glaucoma can develop even under normal pressure. Therefore, lowering the intraocular pressure alone cannot cease optic nerve damage in some patients.

The incidence of POAG is increasing with the aging population. While there were approximately 44 million cases of POAG all over the world in 2013, it was estimated that this number would increase to around 53 million in 2020.

Ethnical differences are very common, and they are more common in the black race than in the white race and Asian race. The prevalence in the black race, where it is most common, was found to be 5.2% at the age of 60 and 12.2% at the age of 80 years. Its incidence increases with age. In some studies, it was observed at similar rates in men and women, while in some studies it was observed slightly more in men.

Family history is a risk factor for POAG. This result reveals the importance of genetic transmission.

Although many risk factors such as high IOP, family history, race, advanced age, and myopia have been identified, the main cause of glaucomatous optic neuropathy is unknown. Humor aqueous (HA), produced by the non-pigmented epithelial cells of the ciliary body, is excreted mostly iridocorneal via the juxtacanalicular trabecular network and Schlemm's canal (conventional), and to a lesser extent by the uveoscleral route and enters the venous circulation. POAG 'Rather, it is known that there is a resistance to conventional outflow at the level of the juxtacanalicular trabecular meshwork and the inner wall of Schlemm's canal. In eyes with glaucoma, histological changes in the collagen structure of the trabecular meshwork, the spaces between the trabecular meshwork, and the juxtacanalicular connective tissue, and changes in endothelial cell functions were detected. In addition to these histological changes, collapse in Schlemm's canal is thought to contribute to the increase in resistance to outflow. Along with these, different theories have been proposed that increase the outflow resistance. These theories can be listed as follows:

* Occlusion of the trabecular meshwork by accumulated substances,
* Loss of trabecular endothelial cells,
* Decreased trabecular mesh pore density in Schlemm canal inner wall endothelium, loss of giant vacuoles,
* Loss of normal phagocytic activity,
* IOP 'Disturbances in the neurological feedback mechanism that concerns the id. In addition, complex mechanisms such as increased oxidative stress, excitotoxicity, hardening of the lamina cribrosa structure, vascular regulation disorder and ischemia, mitochondrial dysfunction, decrease in neurotrophic factors as a result of mechanical stress-induced axoplasmic flow disruption, autoimmunity, low cerebrospinal fluid (CSF) pressure also play a role in the etiopathogenesis.

The aim of the treatment is to preserve the visual functions without impairing the patient's quality of life. When making a treatment plan, the stage of glaucoma, the pressure level at which it progresses, and the expected life expectancy of the patient should be considered.

Life expectancy and the stage of the disease are important criteria in the choice of treatment. A young patient with mild glaucomatous injury should be treated more aggressively than an 80-year-old patient with moderate glaucomatous injury.

Currently, all treatment modalities are aimed at lowering IOP, as IOP is the only factor that can be intervened. According to the treatment protocol accepted all over the world, IOP is tried to be controlled primarily with medical treatment. In cases where medical treatment is insufficient, laser trabeculoplasty or filter surgery is applied.

Today, medical treatment of glaucoma begins with eye drops and usually monotherapy (single molecule therapy). If adequate IOP reduction is not achieved with the drug that is started, it is switched to another drug from the same group. If the target pressure is still not reached, combined therapy is started. In combination therapy, drugs that lower IOP by different mechanisms should be combined. Fixed combinations are preferred for ease of use.

PAAG 'Drugs used in the treatment of:

* Parasympathomimetic drugs (cholinergic drugs),
* Sympathomimetic drugs,
* Beta blockers,
* Hyperosmotic drugs,
* Calcium channel blockers,
* Prostaglandin analogues,
* Carbonic anhydrase inhibitors,
* Rho kinase inhibitors. More than half of patients suffer from progressive visual field loss in long-term medical treatment. However, while the annual rate of visual field loss is 32% in inadequately treated patients, this rate is lower in patients with well-controlled IOP.

These methods are commonly aimed at lowering IOP. However, no method currently used in the clinic can fully treat glaucoma and glaucoma-related neurodegeneration. Unfortunately, despite adequate pressure control, many patients continue to experience irreversible vision loss. The current treatment approach focuses on IOP-independent treatments and neuroprotection.

In this study, flicker light therapy, the effectiveness of which was investigated in the treatment of glaucoma based on some methods used in different diseases, is described for the first time in glaucoma.

In Alzheimer's, another neurodegenerative disease, similar to glaucoma, its pathophysiology is characterized by impaired microcirculation in the brain and retina and pathological chronic activation of microglia, resulting in metabolite accumulation in the extracellular matrix and chronic inflammation, followed by neurodegeneration and axon loss. There are many studies on this subject.

Studies investigating the neurodegenerative properties of glaucoma have found similarities in the pathophysiology of Alzheimer's disease and glaucoma.

40 Hz flicker of light Alzheimer 's the positive effects on the knitted cortex have also been shown in studies. 40 Hz flicker light is aimed to reduce glaucoma and retinal ganglion cell loss due to glaucoma, by reducing neurodegeneration by decreasing amyloid and metabolite accumulation by increasing both microglial phagocytic activation effect and retinal blood flow.

In this study, it was planned to investigate the effect of reducing the progression of glaucomatous damage by applying 40 Hz flicker light therapy for 1 hour a day to POAG patients. It is planned to use visual field test, measurements of retinal nerve fiber layer (RNFL) and ganglion cell complex (GCC) layer thicknesses in optical coherence tomography to investigate the effectiveness of the treatment.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for subject selection

* Those who have applied to the eye diseases clinic
* ≥18 years old
* Those diagnosed with primary open-angle glaucoma (POAG) before the study
* Recipients of standard drug therapy (defined in diagnostic and treatment guidelines) for POAG
* Patients deemed appropriate by the investigator to be included in the study after ophthalmological examination
* According to the results of intraocular pressure (IOP) measurement and visual field test, patients with target pressure and initial moderate visual field loss who were deemed appropriate for inclusion in the study by the investigator
* Patients who were informed about the study and agreed to participate in the study
* Those who agree to continue to use acceptable methods of contraception during the study

Exclusion Criteria:

-

Exclusion criteria for selection of subjects

* Those with a history of trauma or inflammation in their eyes
* Those who have undergone intraocular surgery or laser in the last 6 months, excluding those who have had uncomplicated cataract surgery
* Presence of any retinal or neurological disease other than glaucoma, abnormal ocular motility preventing binocular fixation (eg, nystagmus, strabismus)
* Those with corneal transplants
* Advanced disc cupping (c/d ratio 0.8 and above)
* Large and severe perimetric defects (a central perimetric residual not greater than 10 central degrees)
* Advanced visual field damage (MD above 12 db)
* Dry/wet type age-related macular degeneration in one or both eyes
* Those who have had glaucoma surgery in the past, excluding laser
* Corneal dystrophies
* High myopia (more than 6 diopters)
* Peripheral retinal degenerations with risk of retinal detachment
* Keratitis
* Those with severe dry eye syndrome
* Those with neurological disorders (eg, epilepsy)
* Those with systemic diseases (eg, diabetic mellitus)
* Women who are pregnant supported by biochemical laboratory findings
* Patients with difficulties in understanding and adapting to the study
* Negative benefit/risk ratio determined by the investigator
* Participated in any clinical trial within the previous 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Frequency of the adverse events | 6 months
  In our study, the safety of the GlaucoT glasses with flickering light treatment will be assessed. The purpose of the treatment is to provide neuroprotection with flickering light treatment.
  The primary outcome for safety of the device is the frequency of the adverse events.
The stabilization in visual field test | 6 months
  The second outcome of the clinical trials will be the efficacy of the GlaucoT device. The differences between the patients who use GlaucoT will be compared with the ones that do not use the device under same conditions (e.g. drug use).
  The assessment will be based on visual field test.

CONTACTS AND LOCATIONS:
Overall Officials: Ozcan Kayikcioglu, Prof, Principal Investigator — Manisa Celal Bayar University Department of Ophthalmology
Locations (2):
- Turkey (Türkiye) (2):
  - Ege University Department of Ophthalmology, Izmir
  - Manisa Celal Bayar University Department of Ophthalmology, Manisa

IPD SHARING:
Plan to Share IPD: No
Our clinical research protocol will be shared with other researchers. The results of this clinical study will be published in an academical paper.

REFERENCES:
- [Background] Iaccarino HF, Singer AC, Martorell AJ, Rudenko A, Gao F, Gillingham TZ, Mathys H, Seo J, Kritskiy O, Abdurrob F, Adaikkan C, Canter RG, Rueda R, Brown EN, Boyden ES, Tsai LH. Gamma frequency entrainment attenuates amyloid load and modifies microglia. Nature. 2016 Dec 7;540(7632):230-235. doi: 10.1038/nature20587. PMID 27929004
- [Background] Samanchi R, Prakash Muthukrishnan S, Dada T, Sihota R, Kaur S, Sharma R. Altered spontaneous cortical activity in mild glaucoma: A quantitative EEG study. Neurosci Lett. 2021 Aug 10;759:136036. doi: 10.1016/j.neulet.2021.136036. Epub 2021 Jun 8. PMID 34116196
- See also: The official webpage of the sponsor — http://www.glaucot.com